CLINICAL TRIAL: NCT03679663
Title: Prospective Randomized Controlled Trial to Compare a Handheld Ultrasound Identification of the Neuraxial Block Insertion Site Versus Palpation Only in an Obese Population of Women Undergoing Cesarean Delivery
Brief Title: Ultrasound Versus Palpation for Spinal Anesthesia Success
Acronym: Accuro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TASMC-18-CFW-0219-CTIL
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-01

CONDITIONS: Ultrasound
Keywords: ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Masking Description: The outcomes will be assessed by an observer who was not in the room when the puncture site was identified and was blinded to the study group. The room set up will be identical with the handheld ultrasound placed visible in all cases, including those randomized to the palpation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Palpation (No Intervention): Anesthesia performed without ultrasound
- Ultrasound (Experimental): Anesthesia performed after ultrasound
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Use of ultrasound to identify pre-puncture site
  Arms: Ultrasound

SUMMARY:
Aim is to investigate the difference in number of attempts to place neuraxial block comparing handheld ultrasound versus use of palpation alone for women with impalpable bony landmarks undergoing spinal anesthesia for elective cesarean delivery.

DETAILED DESCRIPTION:
Patients will be recruited prior to cesarean delivery and their site of lumbar injection will be examined. Women with impalpable bony landmarks will be offered recruitment to the study. Women will be randomly assigned to the standard of care group - palpation attempts only, versus an ultrasound group, where the insertion point will be identified by the handheld ultrasound device

Inclusion criteria:

Lumbar spinous processes impalpable. Elective cesarean delivery for singleton pregnancies BMI >30 No contraindications to neuraxial block Signed informed consent Neuraxial Block planned Exclusion Criteria Refuses informed consent Poor written Hebrew, no spoken English or Hebrew Patients will be randomized into two groups : an ultrasound (US) group and a palpation (PP) group.

The primary outcome of our study is the number of needle redirections, defined as any ventral advancement of the needle and/or introducer, as well as any new intervertebral space attempted.

Secondary outcomes include:

The insertion site identification time, patient verbal numerical pain score (0-10) after skin incision.

ELIGIBILITY:
Inclusion Criteria:

Lumbar spinous processes impalpable. Elective caesarean delivery for singleton pregnancies BMI >30 No contraindications to neuraxial block Signed informed consent Neuraxial Block planned

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Needle movement | 10 mins
  number of needle redirections, defined as any ventral advancement of the needle and/or introducer, as well as any new intervertebral space attempted.

SECONDARY OUTCOMES:
The insertion site identification time, | 10 mins
  time
Patient verbal numerical pain score (0-10) after skin incision. | 10 mins
  Patient verbal numerical pain score (0-10) after skin incision. Scale is Verbal numerical rating scale, where zero = no pain at all and 10 = maximum possible pain.
Patient verbal numerical pain score (0-10) after spinal performance. Patient verbal numerical pain score (0-10). Scale is Verbal numerical rating scale, where zero = no pain at all and 10 = maximum possible pain. | 10 mins
  Patient verbal numerical pain score (0-10) after spinal performance. Patient verbal numerical pain score (0-10) Scale is Verbal numerical rating scale, where zero = no pain at all and 10 = maximum possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No